CLINICAL TRIAL: NCT01734707
Title: Atherosclerosis Monitoring and Atherogenicity Reduction Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute for Atherosclerosis Research, Russia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IAR-AMAR
Record Dates: First submitted 2012-11-16; First posted 2012-11-28 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2005-01

CONDITIONS: Carotid Atherosclerosis
Keywords: atherosclerosis; regression; Allicor; garlic; intima-media thickness
MeSH Terms: conditions — Carotid Artery Diseases; Atherosclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- Allicor (Active Comparator): Allicor 150 mg tablet by mouth two times a day
  Interventions: Dietary Supplement: Allicor
- Sugar pill (Placebo Comparator): Placebo tablet 150 mg by mouth two times a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Allicor
  Other Names: time-released garlic powder tablets
  Arms: Allicor
Drug: Placebo — Sugar pill manufactured to mimic Allicor 150 mg tablet
  Arms: Sugar pill

SUMMARY:
This study was designed to estimate the effect of two-year treatment with time-released garlic-based drug Allicor on the progression of carotid atherosclerosis in double-blinded placebo-controlled randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 40 to 74 years
* Subclinical carotid atherosclerosis detected by B-mode ultrasound (increased intima-media thickness 1100-2000 mcm)
* Arterial normotension or mild arterial hypertension (systolic blood pressure <160 mm Hg, diastolic blood pressure <90 mm Hg)
* Absence of chronic diseases demanding permanent drug administration (more than 2 month per year)

Exclusion Criteria:

* Personal history or diagnostic of following diseases:

  1. Transient ischemic attacks
  2. Presence of chronic diseases demanding permanent drug administration (more than 2 month per year)
  3. Condition of patients moderate to severe
* Indications for surgical treatment of atherosclerotic lesions localized in the extracranial brachiocephalic system.
* Individual intolerance of Allicor or appearance of side effects

Ages: 40 Years to 74 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2004-01; Primary Completion 2005-01 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
high-resolution B-mode ultrasonography of common carotid arteries | up to 2 years
  Variation in carotid intima-media thickness (IMT) of the far wall of common carotid arteries

SECONDARY OUTCOMES:
Measure of serum atherogenicity | up to 2 years
  Change of the ability of serum to induce cholesterol accumulation in cultured cells

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Atherosclerosis Research, Moscow, Moscow, Russia

REFERENCES:
- [Result] Sobenin IA, Pryanishnikov VV, Kunnova LM, Rabinovich YA, Martirosyan DM, Orekhov AN. The effects of time-released garlic powder tablets on multifunctional cardiovascular risk in patients with coronary artery disease. Lipids Health Dis. 2010 Oct 19;9:119. doi: 10.1186/1476-511X-9-119. PMID 20958974